CLINICAL TRIAL: NCT07134803
Title: ACCURACY OF ORTHODONTIC BRACKETS POSITIONING WITH OR WITHOUT DENTAL LOUPES
Brief Title: ACCURATE ORTHODONTIC BRACKETS POSITIONING WITH OR WITHOUT DENTAL MAGNIFYING LOUPES
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Joel Moh Heng Shu, University Science Malaysia (USM), Doctor of Dental Surgery. Master of Oral Science (Malaya), University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UMG050E-2024; UMG050E-2024 (Other Grant/Funding Number: FACULTY OF DENTISTRY, UNIVERSITI MALAYA)
Record Dates: First submitted 2025-08-07; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Bracket Bonding; Digital Application; Technology-enhanced Learning
Keywords: Bracket Positioning; Dental Loupes

STUDY DESIGN:
Intervention Model Description: This was a two-arm parallel, singe-centre randomised study where the patients that have been treatment planned were randomised into two groups according to the block pattern:
  Group NL: Bonding of the orthodontic brackets without dental loupe Group L: Bonding of the orthodontic brackets with dental loupe
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group NL: Bonding of the orthodontic brackets without dental loupe (No Intervention): Bonding of the orthodontic brackets on patients' teeth without dental loupe
- Group L: Bonding of the orthodontic brackets with dental loupe (Active Comparator): Bonding of the orthodontic brackets on patients' teeth with dental loupe
  Interventions: Device: Bonding of the orthodontic brackets with dental loupe with Zumax Dental loupes DFK Angled Loupe with a magnification of x3.0 and focus depth of 42cm

INTERVENTIONS:
Device: Bonding of the orthodontic brackets with dental loupe with Zumax Dental loupes DFK Angled Loupe with a magnification of x3.0 and focus depth of 42cm — Bonding of the orthodontic brackets on patients' teeth with dental loupe with Zumax Dental loupes DFK Angled Loupe with a magnification of x3.0 and focus depth of 42cm. Then the scanned for STL file and be superimposed with the gold standard created for the patient individually.
  Arms: Group L: Bonding of the orthodontic brackets with dental loupe

SUMMARY:
The goal of this clinical trial is to assess the accuracy of bracket positioning on tooth facial axis of clinical crown with dental loupes (L) or without dental loupes (NL) on orthodontic patients. The main questions it aims to answer are:

1. Does the usage of dental loupes affect the linear measurement of the bracket positioning during bond-up in patients?
2. Does the usage of the dental loupes affect the angular measurement of the bracket positioning during bond-up in patients ?

Researchers will compare group that use dental loupes and without dental loupes to a gold standard.

Participants will

* Be addressed a treatment plan tailored to their malocclusion.
* Take an intraoral scan with an intraoral scanner 3Shape TRIOS, Copenhagen, Denmark.
* Attend bond up session that was scheduled within a week time once the gold standard for individual patient was generated.
* Take second intraoral scan after bracket bonding

DETAILED DESCRIPTION:
Interventions

This was a two-arm parallel, singe-centre randomised study where the patients that have been treatment planned were randomised into two groups according to the block pattern:

Group NL: Bonding of the orthodontic brackets without dental loupe Group L: Bonding of the orthodontic brackets with dental loupe After extraction procedure was performed according to treatment plan. Within a week, the patient's teeth were dried before taking an intraoral scan with an intraoral scanner 3Shape TRIOS, Copenhagen, Denmark. After scanning the upper and lower arches, the teeth images were stored in STL file. STL file is a format commonly used for 3D printing and computer-aided design (CAD).

The STL file of each patient upper and lower arches were exported and printed into model by the 3D printer by digital dental laboratory to allow extraoral bracket positioning. The extraoral bracket positioning on the twenty 3D printed models were the gold standard for the eighteen patients respectively.

Once the gold standard for individual patient was generated, the bond up session was scheduled within a week time, a new set of brackets were placed by MJHS on the patient's maxillary and mandibular right to left premolars. Bonding of the brackets was performed according to the manufacturer's instructions. Dental loupes Zumax DFK Angled Loupe with a magnification of x3.0 and focus depth of 42cm was used. For the patients bond up by direct eye vision or using dental loupes, the brackets were positioned in the centre of mesial-distal dimension and aligned with the long axis of the crown. No over-correction of the bracket positioning was done to correct specific malocclusions, rotation, or tipping problems. After 40s light-curing of the composite according to manufacturer instructions. The bracket bonding was performed by MJHS in all patients to avoid inter-operator errors.

After bracket bonding, the postoperative dentitions was dried, and scanned with intraoral scanner for T2 by MJHS. Independent assistant (MM) coded the patients scanned STL files which were preoperative (3D images of T1 as gold standard) and postoperative 3D images as a pair without the knowledge of the principal investigator. The software identified 4 identical points on the same teeth from each pair of files and align for superimposition. The different bracket position was shown on the computer's screen in different colours. The differences in mesio-distal (MD) and occlusal-gingival (OG) dimensions, as well as mesio-distal angulation (MDang) dimensions were measured at magnification x10 of superimposition.

To measure the difference in bracket placement between the 2 methods employed the comparison between file preoperative and file postoperative, positive and negative signs were used for distances (distal: +; mesial: -; gingival: +; occlusal: -) and angulation (distal: +; mesial: -). Measurements included all the teeth in the inclusion criteria (Mohammadi & Moslemzadeh, 2011; Panayi et al., 2020).

After the last 0.018" NiTi archwire for full expression of alignment archwire, the patients' teeth again scanned to assess the alignment of the teeth, T3. A crowding score based on the mesio-distal width for the maxillary and mandibular teeth will be measured in millimeters at T3 compared to T2 in relation to the line of arch that reflects the majority of teeth (Kirschen et al., 2000). The alignment of the patients' teeth with be categorized using Little's Irregularity Index into five categories based on a numerical score: 0 indicates perfect alignment, 1-3 is minimal irregularity, 4-6 is moderate irregularity, 7-9 is severe irregularity, and 10 or more is very severe irregularity. This index quantifies the degree of anterior crowding by measuring the sum of linear displacements (mm) of anatomical contact points of six anterior teeth. Any bracket that dislodged from the teeth was bonded back and kept in record. Bracket off was bonded according to the intervention the patient received. The leveling and alignment phase was considered accomplished when 0.019x0.025-inch stainless steel (SS) wire could be inserted without applying an exaggerated force (Al-Ibrahim et al., 2023). The dropout criteria was defined BPE score more than 2.

ELIGIBILITY:
Inclusion Criteria:

* Able to maintain good periodontal health with BPE score 0,1 or 2.
* Healthy teeth without fractures, abrasions, size-shape abnormalities, or poor morphology
* Fully erupted and complete permanent dentition from right to left premolars on maxillary and mandibular arches.
* Overbite and overjet that allowed brackets to be placed on the lower teeth without occlusal interferences.
* Mild and moderate crowding < 8.0 mm.

Exclusion Criteria:

* Patient with craniofacial disorders (e.g. cleft lip and palate, craniofacial syndromes)
* Clinically visible dental caries, proximal restorations (Class II amalgam or composite), build-ups, crowns, onlays that affect the tooth's mesiodistal diameter.
* Patients that required maxillary and mandibular anterior tooth extraction
* Congenital defects or deformed teeth
* Obvious interproximal or occlusal wear of teeth
* Severe crowding (severe overlapping unable to place bracket)
* Infraocclusion, gingival hyperplasia
* Patient that requires sectional mechanics or brackets swapping mechanics in orthodontic treatment.
* Traumatic extraction

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2024-10-02 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
linear measurement (mm) and mesio-distal angulation (degree) dimension on 3D scanned images of brackets position | 2 weeks
  linear measurement (mm) in mesio-distal and occlusal-gingival dimensions
  mesio-distal angulation dimension (degree) on 3D scanned images of brackets position

SECONDARY OUTCOMES:
Alignment of teeth post intervention | up to 6 months
  assess the alignment of patients' maxillary and mandibular teeth from right to left premolars at the end of levelling and aligning stage between with and without dental loupes intervention groups. The alignment of the patients' teeth with be categorized using Little's Irregularity Index into five categories based on a numerical score: 0 indicates perfect alignment, 1-3 is minimal irregularity, 4-6 is moderate irregularity, 7-9 is severe irregularity, and 10 or more is very severe irregularity. This index quantifies the degree of anterior crowding by measuring the sum of linear displacements (mm) of anatomical contact points of six anterior teeth.

CONTACTS AND LOCATIONS:
Overall Officials: Siti Adibah Othman Senior Consultant in Orthodontics, BDS (Malaya), DDS (Bristol), Principal Investigator — Department of Paediatric Dentistry and Orthodontics, Faculty of Dentistry, Universiti Malaya; Roziana Mohd Razi Senior Lecturer & Specialist Orthodontist, BDS (Malaya), MClinDent(Ortho), Principal Investigator — Department of Paediatric Dentistry and Orthodontics, Faculty of Dentistry, Universiti Malaya
Locations (1):
- Department of Paediatric Dentistry and Orthodontics, Faculty of Dentistry, Universiti Malaya, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No
No, we do not plan to share individual participant data (IPD). The dataset will not be made publicly available due to concerns about participant privacy and data sensitivity.